CLINICAL TRIAL: NCT02211118
Title: Sedation and Physiological Effects of Intranasal Dexmedetomidine in Severe COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dayton VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nystrom01
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: COPD; Sedation; Dexmedetomidine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IN-DEX (Experimental): Subjects will be administered 1 mcg/kg or 1.5 mcg/kg intranasal dexemdetomidine (IN-DEX) and monitored for up to 5 hours.
  Interventions: Drug: Intranasal dexemdetomidine (IN-DEX)

INTERVENTIONS:
Drug: Intranasal dexemdetomidine (IN-DEX)
  Other Names: precedex

SUMMARY:
A variety of medications have been used to treat the anxiety, discomfort, and fear associated with continuous and sudden episodic breathlessness in patients with advanced respiratory disease. Opioids and benzodiazepines, used alone or in combination, are commonly prescribed for this distressing symptom. Clinicians are concerned about the adverse effects of opioids, especially respiratory depression, so they frequently prescribe benzodiazepines. Recent studies have shown that benzodiazepine use is associated with increased adverse respiratory outcomes in older adults with Chronic Obstructive Pulmonary Disease (COPD).

Dexmedetomidine may be an alternative to current drug therapies for breathlessness. Dexmedetomidine produces a dose dependent sedation, anxiolysis, and analgesia without respiratory depression or cognitive dysfunction. The drug can be administered intranasally to induce light to moderate sedation of several hours duration.

The objective of the proposed research, a pilot study, is to assess the dose dependent safety and efficacy of intranasal dexmedetomidine in clinically stable patients with severe COPD. This will be accomplished in a staffed acute care setting with routine vital signs monitoring and pulse oximetry. Patients will be assessed objectively and subjectively for their level of sedation by validated sedation scales.

This pilot study is an initial investigation of a drug with favorable pharmacologic properties in this patient population with distressing and difficult to treat symptoms. The pilot study may provide evidence that a larger trial is needed to confirm the study results, or evidence that additional study in symptomatic patients and treatment comparison trials should be pursued.

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD (FEV1 30-50% predicted)
* Age 45-70
* American Society of Anesthesiologists (ASA) Class 3
* Body Mass Index <35 kg/meter squared
* No prior history of adverse reactions to alpha 2 agonists (dexmedetomidine, clonidine)
* Women of non-child bearing age

Exclusion Criteria:

* known adverse reaction, allergy or hypersensitivity, to alpha 2 agonists
* not nothing by mouth (NPO)
* ASA class >3
* Home oxygen therapy >2LPM by nasal cannula continuous use
* Any evidence of nasal mucosal inflammation, irritation, bleeding or ulceration
* Pregnancy, or possibility of pregnancy
* Coronary heart disease with stable or unstable angina
* Baseline heart rate <55 beats per minute
* Bradyarrhythmia, heart block, presence of pacemaker
* Congestive Heart Failure or known Cardiomyopathy (Ejection Fraction <40% by ECHO, MUGA, or myocardial perfusion imaging)
* Cor pulmonale
* Liver disease (hepatic transaminases above the upper limit of normal, cirrhosis, end stage liver disease)
* diagnosis of moderate to severe Obstructive Sleep Apnea
* currently enrolled in any other research study involving drugs or devices

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Modified Observer's Assessment of Alertness/Sedation Scale | every 15 minutes up to 5 hours after intranasal desmedetomidine
Sedation Visual Analog Scale (VAS) | Every 15 minutes up to 5 hours after intranasal dexemdetomidine
Changes in Vital Signs | Every 5 minutes for 90 minutes, then every 15 minutes for up to 5 hours
  Heart rate, noninvasive blood pressure, respitory rate, pulse oximetry

CONTACTS AND LOCATIONS:
Locations (1):
- Dayton VA Medical Center, Dayton, Ohio, United States